CLINICAL TRIAL: NCT04547296
Title: Sodium Bicarbonate Ringer's Solution for Preventing and Treating Hyperlactacidemia During Hepatectomy: a Multicenter, Randomized and Controlled Study
Brief Title: Sodium Bicarbonate Ringer's Solution for Preventing and Treating Hyperlactacidemia During Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Henan Provincial People's Hospital (Other); Henan Cancer Hospital (Other Government); LanZhou University (Other); Affiliated Hospital of Qinghai University (Other); Shaanxi Provincial People's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-071
Record Dates: First submitted 2020-08-25; First posted 2020-09-14 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hyperlactacidemia
Keywords: hyperlactacidemia; Sodium bicarbonate Ringer's solution; Acetate Ringer's solution; hepatectomy
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRS group (Experimental): After entering the operating room, this group were pre-dilated with sodium bicarbonate ringer's solution (30 min, 8 ml/kg), and maintained with 4-5 ml/kg/h sodium bicarbonate ringer's solution during the operation.
  Interventions: Drug: Sodium Bicarbonate Ringer's Solution
- ARS group (Experimental): After entering the operating room, this group were pre-dilated with acetate ringer ringer's solution (30 min, 8 ml/kg), and maintained with 4-5 ml/kg/h acetate ringer's solution during the operation.
  Interventions: Drug: Sodium Bicarbonate Ringer's Solution

INTERVENTIONS:
Drug: Sodium Bicarbonate Ringer's Solution — After the participants enter the operating room, radial artery puncture and catheterization were performed. The blood gas in the non-oxygen state was used as the basic value. A peripheral venous access was established in one upper limb, and the two groups were pre-dilated with sodium bicarbonate Ringer's solution or acetate Ringer's solution (30 min, 8 ml/kg). For laparoscopic surgery, adjust the PaCO2 value to 35-45 mmHg again 10 minutes after the establishment of the pneumoperitoneum. After the operation started, the two groups of participants were maintained with 4-5 ml/kg/h Ringer's solution during the operation. Blood gas was measured every hour after tracheal intubation during the operation, and the last blood gas was measured when the skin was sutured. When the blood gas pH <7.2, 5% sodium bicarbonate injection was given to correct it.
  Other Names: Acetate Ringer's Solution

SUMMARY:
A variety of reasons lead to a sharp increase in lactic acid levels in patients undergoing liver resection, while leading to hyperlactic acidemia, resulting in decreased cardiac output, elevated blood potassium, and response to catecholamines and insulin Damage, increased risk of kidney damage, poor recovery of liver function, decreased immune function, and prolonged hospital stay. Sodium bicarbonate Ringer injection does not contain lactic acid. HCO3- is metabolized by acid-base neutralization in body fluids, and 90% is CO2 The form is excreted from the body by breathing, and only 10% HCO3- is metabolized by the kidney, without the burden of liver metabolism. Physiological concentration of Cl- avoids perchloric acidosis and kidney damage; physiological concentration of Ca2+ and Mg2+ help maintain the body's electrolyte balance and reduce stress-related arrhythmia.The smooth development of this study will help refine the intraoperative fluid management strategy, improve the patient's intraoperative tissue perfusion, maintain the body's acid-base and electrolyte balance, reduce postoperative kidney damage, and improve the patient's quality of life.

DETAILED DESCRIPTION:
This study intends to carry out a high-quality clinical research with design specifications, large sample, multi-center, randomized and controlled methods. From October 9, 2020 to October 9, 2022, participants undergoing hepatectomy surgery under general anesthesia will be recruited. Participants will be randomly assigned, in a 1:1 ratio, to receive Sodium bicarbonate Ringer's solution or control (Acetate Ringer's solution). The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center. After entering the operating room, the two groups were pre-dilated with sodium bicarbonate Ringer or acetate Ringer (30 min, 8 ml/kg). After the operation started, the two groups of participants were maintained with 4-5 ml/kg/h Ringer's solution during the operation. Blood gas index (but are not limited to these data) at intraoperative will be recorded. At the same time, other dates will be recorded.The participation of each patient is scheduled for 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients for selective liver surgery under general anesthesia
2. Age > 18 year，BMI 18 - 40 kg/m2，American society of Anesthesiologists (ASA) grade are between I - III
3. Ability to understand, sign informed consent and cooperate with the intervention and evaluation

Exclusion Criteria:

1. Abnormal renal function：blood creatinine (Cr) and / or urea nitrogen (BUN)> upper limit of normal value; Patients with underlying kidney disease; patients with congenital kidney malformations.
2. In patients with respiratory failure, arterial blood oxygen partial pressure (PaO2) < 60 mmHg, or accompanied by carbon dioxide partial pressure (PaCO2)> 50mmHg; blood oxygen saturation (SpO2) < 90%.
3. A history of myocardial infarction within 6 months before the screening period; history of severe circulatory or respiratory diseases; history of autoimmune diseases; patients with mental illness or neurological disorders that cannot be expressed exactly; patients with a history of epilepsy; patients with pulmonary edema or congestive heart failure.
4. Severe hypercalcemia (Ca2+ > 2.75 mmol/L), hypernatremia (Na+ > 155 mmol/L), hyperkalemia (K+ > 5.5 mmol/L), hyperchloremia (Cl- > 110 mmol/L), Hypermagnesium (Mg2+ > 1.25 mmol/L).
5. Patients with a history of hypothyroidism; pregnant or lactating women.
6. Patients with a history of adverse blood transfusion reactions; those who refuse blood transfusions.
7. Participation in other clinical studies within 3 months before admission to this study.
8. The investigator considers it unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-10-09 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hyperlactacidemia | During the operation
  Diagnostic criteria: Lac ≥ 2 mmol/L, pH ≤ 7.35, HCO3- ≤ 20 mmol/L, PaCO2 <50 mmHg

SECONDARY OUTCOMES:
The incidence of blood gas index disorder | During the operation
  Blood gas was monitored every hour during the operation and the incidence of intraoperative blood gas index disorder was recorded
Incidence of postoperative acute kidney injury | Day 2 after the operation
  The incidence of acute kidney injury within 48h after surgery was recorded
Rate of postoperative complications | Day 30 after the operation
  postoperative complications: cardiovascular complications; pulmonary complications; infection complications; other complications

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, PHD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (7):
- China (7):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Qinghai University Affiliated Hospita, Xining, Qinghai
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang